CLINICAL TRIAL: NCT02881034
Title: Ribavirin Bioavailability After Telaprevir Exposure in Hepatitis C Patients Treated With PEGylated -Interferon/Ribavirin/Telaprevir Triple Therapy
Brief Title: Ribavirin Bioavailability After Telaprevir Exposure
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0557
Record Dates: First submitted 2016-08-18; First posted 2016-08-26 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Hepatitis C
Keywords: Anemia; Antiviral Agents; Glomerular Filtration Rate; Hepatitis C; Ribavirin; Telaprevir
MeSH Terms: conditions — Hepatitis C; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hepatitis C patients: Hepatitis C virus (HCV) infected patients with a previous non-response to pegylated-interferon/ribavirin therapy and re-treated with pegylated-interferon/ribavirin and telaprevir
  Interventions: Drug: Triple therapy

INTERVENTIONS:
Drug: Triple therapy

SUMMARY:
Anemia is more frequent in patients receiving telaprevir with pegylated-interferon/ribavirin than in those receiving pegylated-interferon/ribavirin alone. The objective was to measure the impact of telaprevir on ribavirin bioavailability and to assess the concomitant renal function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hepatitis C virus infection
* Previous non-response to pegylated-interferon/ribavirin therapy
* Re-treatment with pegylated-interferon/ribavirin and telaprevir

Exclusion Criteria:

* Decompensated liver cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatitis C virus (HCV) infected patients with a previous non-response to pegylated-interferon/ribavirin therapy and re-treated with pegylated-interferon/ribavirin and telaprevir
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in ribavirin plasma trough concentration between baseline and week 4 of triple therapy | before telaprevir initiation during the previous course of PEG (pegylated)-IFN (interferon)/ribavirin combination therapy (T-1), and during the early phase (week 4 ± 2 weeks) of therapy
  Plasma ribavirin trough concentrations were measured using a validated high-performance liquid chromatography-diode array detector method, a highly specific, sensible, and precise method of quantification

SECONDARY OUTCOMES:
Change in renal function between baseline and week 4 of triple therapy | Before telaprevir initiation (T-1), and during the early phase (week 4 ± 2 weeks) of therapy
  Renal function was assessed with the commonly used Modification of the Diet in Renal Disease (MDRD) study equation which allows to assess the estimated glomerular filtration rate (eGFR).
Ribavirin plasma trough concentration at week 8 of therapy | at the later phase of therapy (Week 8 ± 2 weeks)
Ribavirin plasma trough concentration after telaprevir withdrawal | after telaprevir cessation (at least 4 weeks after telaprevir withdrawal (Week 16))
Renal function at week 8 of therapy | at the later phase of therapy (Week 8 ± 2 weeks)
Renal function after telaprevir withdrawal | after telaprevir cessation (at least 4 weeks after telaprevir withdrawal (Week 16))

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de la Croix Rousse, Lyon, France